CLINICAL TRIAL: NCT05567835
Title: A Randomized, Open Labeled Phase II Pilot Study of Total Neoadjuvant Chemotherapy With FLOT ( FLOT-TNT) VS Standard Perioperative FLOT ( FLOTPOP) in Patients With Gastric or GEJ Cancer, and Assessment of CTDNA as Correlative Biological Response
Brief Title: A Study of Total Neoadjuvant Chemotherapy With FLOT VS Standard Perioperative FLOT in Patients With Gastric or GEJ Cancer
Acronym: TOGAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Since activation, 3 subjects were enrolled but were not able to be randomized to a treatment arm because of a positive diagnostic laparoscopy result. Given the lack of accrual the study was closed.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Tannaz Armaghnay, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-50068
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric cancer; GEJ cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel

STUDY DESIGN:
Intervention Model Description: This study is a two arm phase II pilot design, with eligible subjects randomized 1:1 to either Arm A ( Investigational arm) or Arm B ( Standard arm). The chemotherapy dose modification will follow routine clinical care. Both arms will receive chemotherapy and curative surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: FLOT-TNT ( Investigational Arm) (Experimental): Arm A is the investigational arm with all 4 cycles of FLOT given as total neoadjuvant chemotherapy prior to surgery. Each cycle is 28 days and consists of 2 chemotherapy sessions given every 14 days. The total number of chemotherapy sessions in Arm A is 8. Every effort will be made to have surgery in week 20 ( -1 to +2 weeks), 4 weeks post C4 on arm A.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Biological: GSCF
- Arm B: FLOT-POP ( Standard Arm) (Experimental): Arm B us the standard perioperative arm with 2 cycles of pre-operative FLOT ( 4 treatment sessions) and 2 cycles ( 4 treatment sessions) of post-operative FLOT. Post-surgery FLOT will start 4-6 weeks post surgery. Each cycle of chemotherapy consists of 28 days and consists of 2 chemotherapy sessions given every 14 days. The total number of chemotherapy sessions in arm B is 8. Every effort should be done to have surgery done in week 12 ( -1 to +2 weeks) post completion of cycle 2 on ARM B.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Biological: GSCF

INTERVENTIONS:
Drug: Fluorouracil — 2600 mg/m2 IV over 26 hours (+/-1 hour) CI with home pump Day 1,15
  Other Names: 5-FU
Drug: Leucovorin — 200 mg mg/m2 IV over 2 hours Day 1,15
  Other Names: LV
Drug: Oxaliplatin — 85 mg/m2 IV over 2 hours Day 1,15
  Other Names: Eloxatin
Drug: Docetaxel — 60 mg/m2 IV over 60 minutes Day 1,15
  Other Names: Taxotere
Biological: GSCF — Recommended on day 2 and 16 of C1 of the protocol while getting chemotherapy Day 2,16

SUMMARY:
This is a randomized pilot study to evaluate and to compare the completion rates of Total Neoadjuvant chemotherapy with FLOT ( FLOT-TNT) and perioperative chemotherapy with FLOT ( FLOT-POP).

DETAILED DESCRIPTION:
Participants will be randomized 1:1 to either total Neoadjuvant chemotherapy with with FLOT-TNT ( all 4 cycles of chemotherapy before surgery) or standard of care FLOT-POP ( 2 cycles of chemotherapy before surgery and 2 cycles of chemotherapy after surgery). Each cycle of chemo is 28 days long with chemo administered on Days 1 and Day 15 of the cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent.
2. Must be ≥18 years of age.
3. Must have life expectancy of greater than 3 months.
4. Must have pathologically proven Siewert type II or III GEJ or gastric adenocarcinoma from the main tumor or local lymph nodes (pre-neoadjuvant chemo).
5. Stage cT2 or higher, any N and M0, are eligible for the study.
6. M0 disease must be established by both negative distant metastatic disease on imaging AND negative diagnostic laparoscopic assisted cytology of peritoneal fluid cytology not more than 42 days before registration.
7. Must be a candidate for neoadjuvant chemotherapy.
8. Must be a candidate for curative surgical approach.
9. Must have an ECOG performance status 0-2.
10. Male or female subjects of childbearing potential must be willing to use contraceptive precautions throughout the trial and for 3 months after discontinuation of study treatment. Female subjects of childbearing potential must have a negative pregnancy test within 28 days of registration. Post-menopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential.
11. Must have adequate kidney, liver, and bone marrow function, within 28 days prior to registration, as follows:

i. Hemoglobin ≥ 8.0 gm/dL (PRBC transfusion is allowed to meet this criteria) ii. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 iii. Platelet count ≥ 100,000 /mm3 iv. Total bilirubin ≤ 1.5 times upper limit of normal (ULN) v. AST (SGOT) and ALT (SGPT) ≤ 3.0 times the ULN vi. Patient must have adequate renal function as evidenced by one of the following: Serum creatinine ≤ IULN OR calculated creatinine clearance ≥ 60 mL/min. This serum creatinine result must be obtained within 28 days prior to registration.

l. Subjects who have required a short course urgent single modality non curative radiation treatment or gastric artery embolization for the purpose of tumor bleeding control are eligible.

Exclusion Criteria:

1. Positive cytology or histology for metastatic disease on diagnostic laparoscopy peritoneal fluid. Reports such as: "cannot rule out malignancy" or "suspicious for malignancy, but not definitive" will exclude the subject from enrolling.
2. Seiwert type I GEJ cancer
3. Subjects with clinical evidence of metastatic disease.
4. Biopsy proven metastatic disease (excluding regional lymph nodes)
5. Prior chemotherapy for gastric cancer or GEJ cancer
6. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, current non-advanced prostate cancer per the discretion of the investigator, and any other cancers from which the patient has been disease free for two years.
7. Female subjects who are pregnant, breast feeding, or of childbearing potential with a positive pregnancy test prior to baseline. Women of childbearing potential must have a negative serum pregnancy test as a part of eligibility within 28 days of registration. A persistent positive or elevated urine or blood Beta HCG test may be contributed to the primary diagnosis of GC or GEJ cancer after ruling out ectopic and intrauterine pregnancy and germ cell tumors.
8. Subjects unwilling or unable to comply with the protocol or provide written informed consent.
9. Any medical condition that, in the opinion of the investigator, would exclude the subject from participating in this study and treatment plan.
10. ECOG > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Completion rate of Participants who have completed their all-allocated treatments, either Arm A: FLOT-TNT or Arm B: FLOT-POP | at week 16 for Arm A and at week 24 for Arm B
  ArmA has all 4 cycles of FLOT given prior to surgery and ArmB has 2 cycles of pre-operative FLOT and 2 cycles of post-operative FLOT. Each cycle consists of 28 days and consists of 2 chemotherapy sessions given every 14 days. The completion rate of participants is presented based on the number of participants who have completed all treatments by their arms.

SECONDARY OUTCOMES:
Pathologic response rate | at week 12 for Arm A and at week 20 for Arm B
  The pathological response will be evaluated by using Mandard tumor regression grade (TRG) in the primary tumor. Mandard TRG score is from TRG0 (complete response), TRG1 (near-complete response), TRG2 (partial response), and TRG3 (poor or no response).
Number of positive lymph nodes | at week 12 for Arm A and at week 20 for Arm B
  Nodal status is assessed as positive or negative on pathology. The number of positive lymph nodes is obtained from post gastrectomy surgical specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Tannaz Armaghany, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - Baylor College of Medicine Medical Center - McNair Campus, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Ben Taub Hospital, Houston, Texas
  - Harris Health System- Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No